**Informed Consent** 

**Project Name**: Intervention study on self-care ability of patients with rectal cancer

after permanent colostomy

Project leader: Shali Wen

You will be invited to participate in an intervention study on the self-care ability of

patients with permanent colostomy after rectal cancer.

The purpose of this project is to understand the status of ostomy-related

self-efficacy and ostomy self-care and self-esteem in patients with early rectal cancer

after colostomy; and to compile the intervention manual "We can do the same –

enterostomy self-care management" and corresponding Evaluation tool; explores

self-care management (change stage, perceived benefit, perceived disorder, change

process, self-efficacy) and stoma-related self-efficacy, ostomy self-care for patients

with rectal cancer colostomy based on cross-theoretical model (TTM) intervention

model The impact of skills, self-esteem, and quality of life.

This project will be investigated by a professional who has obtained a nurse

qualification.

The project will start on August 1, 2012 to March 31, 2013. It will take 7 months. If

you agree to participate in this program, you will be asked to fill out the

questionnaire.

**Compensation/cost:** There will be no cost to participate in this study. We will give

you a gift cost 10 to 15 yuan as a compensation for participating in this study.

**Risk:** Participation in this study does not result in known physical harm.

Confidentiality: The information you provide will be kept strictly confidential (your name will not be recorded or appear on other research materials). We will number your information and any information that identifies you will be blocked. Your name will not appear when the research results are presented.

**Voluntary participation:** You are free to choose to participate or not to participate. If you participate, you can withdraw at any time for any reason without affecting the services provided by your community.

**Question:** Regarding this research project, if you have any questions, you can ask now. If you have any questions in the future, please call 86-18874751685 to Shali Wen. If you have any questions concerning the protection of the rights of the research object, please contact the Medical Ethics Review Committee of the Second Xiangya Hospital of Central South University, telephone number 86-0731-84896038.

I have read the content provided above and I have been told about the risks and inconveniences and possible benefits of participating in this project. I was also told about the measures I can take in addition to the measures provided by the project. I understand that I can not participate in this project. If I refuse to participate, I will not have any punishment or influence my rights. I can also quit this project at any time.

I understand the rights I should enjoy as a research subject. I am volunteered to participate in this study. I understand what this research is doing, why do you want to do this research and what to do. I will receive a signed informed consent form.

Signature of participant:

day/ month /year

Signature of project leader: Shali Wen

Phone number: 86-18874751685